CLINICAL TRIAL: NCT00775866
Title: MRI - Guided Biopsy for Suspicion of Locally Recurrent Prostate Cancer After External Beam Radiotherapy
Brief Title: MRI-Guided Biopsy of Recurrent Prostate Cancer After Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 05-0641-C; Proposal Number PC050204; Award Number W81XWH-05-1-0570
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Recurrent Prostate Cancer
Keywords: prostate cancer, magnetic resonance imaging, guided imagery
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRI guided prostate biopsy (Experimental)
  Interventions: Procedure: MRI-Guided Biopsy

INTERVENTIONS:
Procedure: MRI-Guided Biopsy — Technical development and clinical testing of a novel technique for magnetic resonance imaging (MRI) guided prostate biopsy in a 1.5T horizontal bore scanner using a dedicated interventional table.

SUMMARY:
In this study we will test a new procedure to guide needle biopsies into the prostate gland based on MRI. This study will be conducted in patients who may have recurrence of their cancer in the prostate gland after radiation therapy in order to map out the location of the recurrence. Using this technique, we will be able to measure the accuracy of MR images in identifying the site of tumour recurrence.

DETAILED DESCRIPTION:
This study involves the technical development and clinical testing of a novel technique for magnetic resonance imaging (MRI) guided prostate biopsy in a 1.5T horizontal bore scanner using a dedicated interventional table. We primarily hypothesize that the integration of diagnostic and interventional MRI enables needle biopsy targeting to foci of tumor recurrence after radiotherapy, and will enable a determination of the diagnostic accuracy of MRI in mapping sub-sites of tumor recurrence after radiotherapy. RELEVANCE TO PUBLIC HEALTH: Patients with recurrence of their prostate cancer after radiotherapy currently face difficult choices. Standard second line treatments target the entire prostate gland and are associated many side effects. This study will directly improve the detection, spatial delineation, and characterization of prostate cancer persistence after radiotherapy. If anatomic patterns of disease persistence are found across patients, radiation delivery techniques will be suitably modified, which may translate to improved cure rates. Importantly, this study will establish a procedural platform for MRI-guidance of minimally invasive local salvage therapies. By precisely focusing salvage therapy to sites of tumor persistence within the prostate gland, side effects may be reduced in the future.

ELIGIBILITY:
Inclusion Criteria:

* Biochemical failure > 18 months after definitive external beam radiotherapy (ASTRO definition - revised version 2006: rise by 2 ng/mL or more above the nadir PSA)
* PSA <20 prior to initial course of external beam radiotherapy
* PSADT >3 months at failure
* Age ≥ 18 years
* ECOG performance status 0 or 1 with >10 year life expectancy
* Fit for local anaesthesia
* Informed consent:

Exclusion Criteria:

* Contraindications to MRI
* Severe claustrophobia
* Bleeding diathesis and anti-coagulative therapy that cannot be temporarily ceased precluding brachytherapy
* Previous brachytherapy
* Active hormonal therapy
* Radiologic evidence of LN or distant metastases
* Other urinary or medical conditions deemed by the PI or associates to make the patient ineligible for MRI-guided prostate biopsy.
* Contraindications to endorectal coil, surgically absent rectum, severe hemorrhoids or previous colorectal surgery
* Contraindications to conscious sedation
* Contraindication to IV Gadolinium administration
* latex allergy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2006-10; Primary Completion 2015-05 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is a preliminary estimate of the diagnostic accuracy of MRI in identifying sites of recurrent tumor after radiotherapy for prostate cancer. | at the end of the evaluation phase

CONTACTS AND LOCATIONS:
Overall Officials: Peter Chung, MB ChB, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Menard C, Iupati D, Publicover J, Lee J, Abed J, O'Leary G, Simeonov A, Foltz WD, Milosevic M, Catton C, Morton G, Bristow R, Bayley A, Atenafu EG, Evans AJ, Jaffray DA, Chung P, Brock KK, Haider MA. MR-guided prostate biopsy for planning of focal salvage after radiation therapy. Radiology. 2015 Jan;274(1):181-91. doi: 10.1148/radiol.14122681. Epub 2014 Sep 8. PMID 25203127